CLINICAL TRIAL: NCT06474975
Title: SURGYPET: Intra-SURGerY High-resolution Specimen PET/CT Imager for Margin Assessment in Early-stage Breast Cancer as Compared to Gross Pathology: a Prospective Non-inferiority Analysis
Brief Title: Intra-SURGerY High-resolution Specimen PET/CT Imager for Margin Assessment in Early-stage Breast Cancer
Acronym: SURGYPET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: L2-092
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Breast-conserving Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Identification of positive margins with PET/CT specimen imager (Experimental): Identification of all positive margins of the invasive component during BCS using PET/CT specimen imager
  Interventions: Device: AURA 10 PET/CT

INTERVENTIONS:
Device: AURA 10 PET/CT — The PET/CT specimen imager (AURA 10 PET/CT) is used to intraoperatively assess resection margins and histopathological findings of the breast tumor specimen are applied as the gold standard
  Other Names: PET/CT specimen imager (AURA 10 PET/CT)

SUMMARY:
This study is a diagnostic open-label, prospective, single-arm non-inferiority clinical trial.

The primary endpoint is the accuracy to detect positive invasive margins in invasive ductal carcinoma (IDC) patients by high-resolution specimen Positron Emission Tomography/Computed Tomography (PET/CT) imaging.

DETAILED DESCRIPTION:
The rationale of this study is to examine the non-inferiority of intraoperative high-resolution specimen PET/CT imaging in early-stage breast cancer for the identification of all positive margins of the invasive component during Breast Cancer Surgery (BCS) as compared to standard-of-care gross pathology evaluation.

The PET/CT specimen imager is used to intraoperatively assess resection margins and histopathological findings of the breast tumor specimen are applied as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* females with an age over 18 years;
* confirmed breast cancer with indication to undergo BCS (stage I-II with tumor ≤2.5 in greatest dimension);
* vacuum-assisted core breast biopsy is allowed for non-invasive tumors only;
* able to understand treatment protocol and informed consent form;
* estimated by the investigator to be compliant for study participation.

Exclusion Criteria:

* general or local contra-indication for BCS;
* previous breast surgery;
* inflammatory breast cancer;
* radiotherapy of the ipsilateral breast;
* vacuum-assisted core breast biopsy for all patients with invasive tumors (vacuum-assisted core breast biopsy is allowed for patients with non-invasive tumors as long as the residual tumor size on mammogram is at least 1.0 cm);
* pregnancy or lactation;
* participation in other clinical studies with a radiation exposure of more than 1 mSv in the past year;
* active bacterial, viral or fungal infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the accuracy to detect positive invasive margins in IDC patients | 1 month
  Evaluation of intraoperative high-resolution specimen PET/CT imaging for the identification of all invasive positive margins during primary breast-conserving surgery (BCS) of invasive ductal carcinoma (IDC), as compared to perioperative gross pathology evaluation. Permanent pathology is used as the gold standard for margin assessment.

SECONDARY OUTCOMES:
Evaluation of diagnostic performance of PET/CT in the detection of positive margins respect to gross pathology | 1 month
  determining the diagnostic performance of intraoperative high-resolution specimen PET/CT imaging and gross pathology to detect all positive margin;
Detection of malignant cells in resected lymph nodes and cavity shaves | 1 month
  exploring the ability of intraoperative high-resolution specimen PET/CT imaging to detect the presence of malignant cells in resected lymph nodes and cavity shaves;
Definition of optimal SUVmax cut-off | 1 months
  determining the optimal SUVmax cut-off in intraoperative high-resolution specimen PET/CT imaging for the correct detection of malignant vs. non-malignant tissues, using pathology results as standard-of-reference

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Ceci, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy